CLINICAL TRIAL: NCT00002996
Title: Flecainide for the Treatment of Chronic Neuropathic Pain: A Phase II Trial
Brief Title: Flecainide in Treating Patients With Chronic Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Purpose: Supportive Care
Other Study IDs: CDR0000065544; E1Z95
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: flecainide acetate

SUMMARY:
RATIONALE: Flecainide therapy may help patients with neuropathic pain live more comfortably.

PURPOSE: Phase II trial to study the effectiveness of flecainide in treating patients with chronic neuropathic pain from cancer or AIDS.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate the effectiveness of flecainide in the management of neuropathic pain.

OUTLINE: Patients are given a brief pain inventory (BPI) form to assess their pain upon enrollment in the study. Following a 7 day stabilization period, flecainide is administered. One capsule of flecainide is given twice a day on days 8-10, two capsules are given twice a day on days 11-14 and three capsules are given twice a day on days 15-21. BPI forms are completed on days 8, 15 and 22 to assess neuropathic pain.

PROJECTED ACCRUAL: A total of 7-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Chronic neuropathic pain with diagnosis of cancer or AIDS

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* SGOT no greater than 2 times upper limit of normal (ULN)

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No clinical history of infarction or angina
* No advanced heart failure
* No sick sinus syndrome, intraventricular conduction disease, second or third degree AV block or arrhythmias requiring treatment (exception may be granted by cardiac consult)
* No focal wall motion abnormalities
* Ejection fraction at least 40%
* Systolic blood pressure at least 90 mm Hg

Other:

* Must be able to take oral medication
* No known allergy or adverse reaction to flecainide, mexilitene or any other type I antiarrhythmic drug
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 weeks since prior chemotherapy that may cause neuropathy

Endocrine therapy:

* At least 2 weeks since prior corticosteroids

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No tricyclic antidepressant treatment within past 2 weeks
* No concurrent use of flecainide, mexiletene or any other type I antiarrhythmic drug

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-05-04 (Actual); Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles F. Von Gunten, MD, PhD, Study Chair — Robert H. Lurie Cancer Center
Locations (6):
- United States (6):
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] von Gunten CF, Eappen S, Cleary JF, Taylor SG 4th, Moots P, Regevik N, Cleeland C, Cella D. Flecainide for the treatment of chronic neuropathic pain: a Phase II trial. Palliat Med. 2007 Dec;21(8):667-72. doi: 10.1177/0269216307083031. PMID 18073252